CLINICAL TRIAL: NCT00614393
Title: A Phase II/III Study of Dalotuzumab (MK-0646) Treatment in Combination With Cetuximab and Irinotecan for Patients With Metastatic Colorectal Cancer
Brief Title: Study of Dalotuzumab (MK-0646) in Combination With Cetuximab and Irinotecan in Metastatic Colorectal Cancer (MK-0646-004)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0646-004; 2007_529 (Other: Telerex Number)
Record Dates: First submitted 2008-01-17; First posted 2008-02-13 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — dalotuzumab; Irinotecan; Cetuximab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Dalotuzumab 10 mg/kg Q1W (DB) (Experimental): In double-blind (DB) Week 1, participants receive cetuximab 400 mg/m^2 intravenously (IV) loading dose and irinotecan IV at their pre-study dosage. Starting with DB Week 2, participants receive cetuximab 250 mg/m^2 IV one time each week (Q1W) maintenance dose, irinotecan IV Q1W and DB dalotuzumab 10 mg/kg IV Q1W for up to 32 months of treatment.
  Interventions: Biological: dalotuzumab; Drug: irinotecan hydrochloride; Biological: cetuximab
- Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (OL) (Experimental): In the open-label (OL) portion of the study, ≥6 participants receive cetuximab 400 mg/m^2 Q1W + irinotecan Q1W at their pre-study dosage + OL dalotuzumab (loading dose of 15 mg/kg IV followed by a maintenance dose of 7.5 mg/kg 2 weeks later) to verify the safety of the regimen. In DB Week 1, participants receive cetuximab 400 mg/m^2 IV + irinotecan IV. In DB Week 2, participants receive cetuximab 250 mg/m^2 IV + irinotecan IV + DB dalotuzumab 15 mg/kg IV. In DB Week 3, participants receive cetuximab 250 mg/m^2 IV + irinotecan IV. Starting with DB Week 4, participants receive cetuximab 250 mg/m^2 IV Q1W + irinotecan IV Q1W + DB dalotuzumab 7.5 mg/kg IV Q2W for up to 32 months of treatment.
  Interventions: Biological: dalotuzumab; Drug: irinotecan hydrochloride; Biological: cetuximab
- Dalotuzumab 10 mg/kg Q1W (OL) (Experimental): In the OL portion of the study, ≥6 participants receive cetuximab 400 mg/m^2 Q1W+ irinotecan Q1W at their pre-study dosage + OL dalotuzumab 10 mg/kg IV Q1W to verify the safety of the regimen. In DB Week 1, participants receive cetuximab 400 mg/m^2 IV + irinotecan IV at their pre-study dosage. Starting with DB Week 2, participants receive cetuximab 250 mg/m^2 IV Q1W + irinotecan IV Q1W + DB dalotuzumab 10 mg/kg IV Q1W for up to 32 months of treatment.
  Interventions: Biological: dalotuzumab; Drug: irinotecan hydrochloride; Biological: cetuximab
- Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (DB) (Experimental): In DB Week 1, participants receive cetuximab 400 mg/m^2 IV + irinotecan IV at their pre-study dosage. In DB Week 2, participants receive cetuximab 250 mg/m^2 IV + irinotecan IV + DB dalotuzumab 15 mg/kg IV. In DB Week 3, participants receive cetuximab 250 mg/m^2 IV + irinotecan IV. Starting with DB Week 4, participants receive cetuximab 250 mg/m^2 IV Q1W + irinotecan IV Q1W + DB dalotuzumab 7.5 mg/kg IV Q2W for up to 32 months of treatment.
  Interventions: Biological: dalotuzumab; Drug: irinotecan hydrochloride; Biological: cetuximab
- Placebo + Cetuximab + Irinotecan (DB) (Active Comparator): In DB Week 1, participants receive cetuximab 400 mg/m^2 IV + irinotecan IV at their pre-study dosage. Starting with DB Week 2, participants receive cetuximab 250 mg/m^2 IV Q1W + irinotecan IV Q1W + DB normal saline (placebo) IV Q1W for up to 32 months of treatment.
  Interventions: Drug: irinotecan hydrochloride; Biological: cetuximab; Drug: placebo

INTERVENTIONS:
Biological: dalotuzumab — IV infusion
  Other Names: MK-0646
  Arms: Dalotuzumab 10 mg/kg Q1W (DB); Dalotuzumab 10 mg/kg Q1W (OL); Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (DB); Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (OL)
Drug: irinotecan hydrochloride — IV infusion
  Other Names: CAMPTOSAR®
Biological: cetuximab — IV infusion
  Other Names: ERBITUX®
Drug: placebo — IV infusion
  Other Names: placebo to dalotuzumab; normal saline solution
  Arms: Placebo + Cetuximab + Irinotecan (DB)

SUMMARY:
This study will compare the safety and efficacy of dalotuzumab (MK-0646) in combination with cetuximab and irinotecan in treating participants with wild type KRAS (wtKRAS) metastatic colorectal cancer (CRC) compared to cetuximab and irinotecan alone.

The primary study hypothesis is that administration of dalotuzumab in combination with cetuximab and irinotecan to participants with metastatic CRC expressing the wtKRAS genotype improves Overall Survival OR Progression-free Survival compared to participants treated with cetuximab and irinotecan alone.

DETAILED DESCRIPTION:
Dalotuzumab is a humanized monoclonal antibody (mAb) that targets the insulin-like growth factor type 1 receptor-1 (IGF-1R). Dalotuzumab may act through inhibition of insulin-like growth factor-1 (IGF-1)-mediated cell signaling to cause reductions in tumor growth and spread antibody dependent cell-mediated cytotoxicity.

In preclinical studies, dalotuzumab improved the activity of an anti-epidermal growth factor receptor (EGFR) mAb and the activity of erlotinib, a small molecule inhibitor of EGFR.

All eligible participants will receive cetuximab 400 mg/m^2 infusion over 120 minutes followed by weekly infusions of cetuximab 250 mg/m^2 over 60-120 minutes along with irinotecan infusion over 30-90 minutes. Dosage of irinotecan will be the same as most recent pre-study therapy. Participants will then be assigned to one of three treatment double-blind arms.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have confirmed wtKRAS CRC.
* Participant must have previously failed both irinotecan and oxaliplatin containing regimens, and should have progressed on or within 3 months of completing their last line of therapy with objective evidence of progression as verified by previous radiologic scans.

Exclusion Criteria:

* Participant has had cancer treatment within 2 weeks before the first dose of study drug(s) or if the side effects from the drugs have not gone down to a certain level 2 weeks before the first dose of study drugs.
* Participant has had a bad side effect to irinotecan therapy.
* Participant has human immunodeficiency virus (HIV).
* Participant has Hepatitis B or C.
* Participant is pregnant or breast feeding or planning to have a child while on this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2007-12-24 (Actual); Primary Completion 2010-06-01 (Actual); Study Completion 2012-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Sclafani F, Kim TY, Cunningham D, Kim TW, Tabernero J, Schmoll HJ, Roh JK, Kim SY, Park YS, Guren TK, Hawkes E, Clarke SJ, Ferry D, Frodin JE, Ayers M, Nebozhyn M, Peckitt C, Loboda A, Mauro DJ, Watkins DJ. A Randomized Phase II/III Study of Dalotuzumab in Combination With Cetuximab and Irinotecan in Chemorefractory, KRAS Wild-Type, Metastatic Colorectal Cancer. J Natl Cancer Inst. 2015 Sep 23;107(12):djv258. doi: 10.1093/jnci/djv258. Print 2015 Dec. PMID 26405092

RESULTS

PARTICIPANT FLOW:
Groups:
- Dalotuzumab 10 mg/kg Q1W (DB): In double-blind (DB) Week 1, participants received cetuximab 400 mg/m^2 intravenously (IV) loading dose and irinotecan IV at their pre-study dosage. Starting with DB Week 2, participants received cetuximab 250 mg/m^2 IV one time each week (Q1W) maintenance dose, irinotecan IV Q1W and DB dalotuzumab 10 mg/kg IV Q1W for up to 32 months of treatment.
- Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (OL): In the open-label (OL) portion of the study, ≥6 participants received cetuximab 400 mg/m^2 Q1W + irinotecan Q1W at their pre-study dosage + OL dalotuzumab (loading dose of 15 mg/kg IV followed by a maintenance dose of 7.5 mg/kg 2 weeks later) to verify the safety of the regimen. In DB Week 1, participants received cetuximab 400 mg/m^2 IV + irinotecan IV. In DB Week 2, participants received cetuximab 250 mg/m^2 IV + irinotecan IV + DB dalotuzumab 15 mg/kg IV. In DB Week 3, participants received cetuximab 250 mg/m^2 IV + irinotecan IV. Starting with DB Week 4, participants received cetuximab 250 mg/m^2 IV Q1W + irinotecan IV Q1W + DB dalotuzumab 7.5 mg/kg IV one time every two weeks (Q2W) for up to 32 months of treatment.
- Dalotuzumab 10 mg/kg Q1W (OL): In the OL portion of the study, ≥6 participants received cetuximab 400 mg/m^2 Q1W+ irinotecan Q1W at their pre-study dosage + OL dalotuzumab 10 mg/kg IV Q1W to verify the safety of the regimen. In DB Week 1, participants received cetuximab 400 mg/m^2 IV + irinotecan IV at their pre-study dosage. Starting with DB Week 2, participants received cetuximab 250 mg/m^2 IV Q1W + irinotecan IV Q1W + DB dalotuzumab 10 mg/kg IV Q1W for up to 32 months of treatment.
- Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (DB): In DB Week 1, participants received cetuximab 400 mg/m^2 IV + irinotecan IV at their pre-study dosage. In DB Week 2, participants received cetuximab 250 mg/m^2 IV + irinotecan IV + DB dalotuzumab 15 mg/kg IV. In DB Week 3, participants received cetuximab 250 mg/m^2 IV + irinotecan IV. Starting with DB Week 4, participants received cetuximab 250 mg/m^2 IV Q1W + irinotecan IV Q1W + DB dalotuzumab 7.5 mg/kg IV Q2W for up to 32 months of treatment.
- Placebo + Cetuximab + Irinotecan (DB): In DB Week 1, participants received a cetuximab 400 mg/m^2 IV + irinotecan IV at their pre-study dosage. Starting with DB Week 2, participants received cetuximab 250 mg/m^2 IV Q1W + irinotecan IV Q1W + DB normal saline (placebo) IV Q1W for up to 32 months of treatment.
Period: Overall Study
Arm/Group | Dalotuzumab 10 mg/kg Q1W (DB) | Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (OL) | Dalotuzumab 10 mg/kg Q1W (OL) | Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (DB) | Placebo + Cetuximab + Irinotecan (DB)
Started | 180 | 8 | 10 | 180 | 180
Treated | 180 | 8 | 10 | 180 | 178
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 180 | 8 | 10 | 180 | 180
Not completed — Adverse Event | 20 | 2 | 3 | 13 | 21
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 2
Not completed — Physician Decision | 17 | 0 | 1 | 8 | 9
Not completed — Progressive Disease | 118 | 5 | 5 | 138 | 130
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0
Not completed — Terminated by Sponsor | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 20 | 1 | 1 | 16 | 13
Not completed — Other | 4 | 0 | 0 | 4 | 2
Not completed — Not Treated | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population was the All Participants As Treated (APAT) population and consisted of all participants who received at least one dose of study drug.
Groups:
- Dalotuzumab 10 mg/kg Q1W (DB): In DB Week 1, participants received cetuximab 400 mg/m^2 IV loading dose and irinotecan IV at their pre-study dosage. Starting with DB Week 2, participants received cetuximab 250 mg/m^2 IV Q1W maintenance dose, irinotecan IV Q1W and DB dalotuzumab 10 mg/kg IV Q1W for up to 32 months of treatment.
- Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (OL): In the OL portion of the study, ≥6 participants received cetuximab 400 mg/m^2 Q1W + irinotecan Q1W at their pre-study dosage + OL dalotuzumab (loading dose of 15 mg/kg IV followed by a maintenance dose of 7.5 mg/kg 2 weeks later) to verify the safety of the regimen. In DB Week 1, participants received cetuximab 400 mg/m^2 IV + irinotecan IV. In DB Week 2, participants received cetuximab 250 mg/m^2 IV + irinotecan IV + DB dalotuzumab 15 mg/kg IV. In DB Week 3, participants received cetuximab 250 mg/m^2 IV + irinotecan IV. Starting with DB Week 4, participants received cetuximab 250 mg/m^2 IV Q1W + irinotecan IV Q1W + DB dalotuzumab 7.5 mg/kg IV Q2W for up to 32 months of treatment.
- Placebo + Cetuximab + Irinotecan (DB): In DB Week 1, participants received cetuximab 400 mg/m^2 IV + irinotecan IV at their pre-study dosage. Starting with DB Week 2, participants received cetuximab 250 mg/m^2 IV Q1W + irinotecan IV Q1W + DB normal saline (placebo) IV Q1W for up to 32 months of treatment.
- Total: Total of all reporting groups
Arm/Group | Dalotuzumab 10 mg/kg Q1W (DB) | Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (OL) | Dalotuzumab 10 mg/kg Q1W (OL) | Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (DB) | Placebo + Cetuximab + Irinotecan (DB) | Total
Number analyzed (Participants) | 180 | 8 | 10 | 180 | 178 | 556
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.6 (10.2) | 55.6 (16.1) | 64.4 (8.9) | 59.4 (10.9) | 58.4 (11.1) | 59.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 3 | 3 | 70 | 62 | 192
  Male | 126 | 5 | 7 | 110 | 116 | 364

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: The OS of participants with metastatic colorectal cancer (CRC) expressing the KRAS wild-type (wtKRAS) tumor genotype (indicating no detection of KRAS mutation) was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. OS was analyzed using the Kaplan-Meier method and is reported in months.
Time Frame: Up to 12 weeks after last dose of study drug (Up to 35 months)
Population: The Intent-to-Treat (ITT) population consisted of all participants who had a wtKRAS tumor genotype. The efficacy analyses were planned for and only included participants from the DB portion of the study. Participants from the OL portion were excluded from the analyses. Participants were counted in the group to which they were randomized.
Measure: Median (Full Range); unit: Months
Arm/Group | Dalotuzumab 10 mg/kg Q1W (DB) | Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (OL) | Dalotuzumab 10 mg/kg Q1W (OL) | Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (DB) | Placebo + Cetuximab + Irinotecan (DB)
Number analyzed (Participants) | 116 | 0 | 0 | 117 | 111
Months | 10.8 [7.9 to 12.9] |  |  | 11.6 [9.6 to 14.3] | 14.0 [10.7 to 16.1]
Statistical Analysis 1: Comparison: Dalotuzumab 10 mg/kg Q1W (DB) vs Placebo + Cetuximab + Irinotecan (DB); Test type: Superiority or Other; p = 0.06, Regression, Cox; Hazard Ratio (HR) = 1.41, 95% CI 2-sided [0.99 to 2.00]
Statistical Analysis 2: Comparison: Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (DB) vs Placebo + Cetuximab + Irinotecan (DB); Test type: Superiority or Other; p = 0.18, Regression, Cox; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [0.89 to 1.79]

2. Primary Outcome: Progression-free Survival (PFS)
Description: The PFS of participants with metastatic CRC expressing the wtKRAS genotype was defined as the time from the first day of study treatment to the first documented disease progression per Response Evaluation Criteria in Solid Tumors version 1.0 (RECIST 1.0) as documented by an independent core laboratory, or death due to any cause, whichever occurred first. Disease progression was defined as either a 20% or greater relative increase in the sum of diameters of target lesions OR an absolute increase of at least 5mm in the sum of lesions or the appearance of new lesions. PFS was analyzed using the Kaplan-Meier method and is reported in months.
Time Frame: Up to last dose of study drug (Up to 32 months)
Population: The ITT population consisted of all participants who had a wtKRAS tumor genotype. The efficacy analyses were planned for and only included participants from the DB portion of the study. Participants from the OL portion were excluded from the analyses. Participants were counted in the group to which they were randomized.
Measure: Median (Full Range); unit: Months
Arm/Group | Dalotuzumab 10 mg/kg Q1W (DB) | Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (OL) | Dalotuzumab 10 mg/kg Q1W (OL) | Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (DB) | Placebo + Cetuximab + Irinotecan (DB)
Number analyzed (Participants) | 116 | 0 | 0 | 117 | 111
Months | 3.9 [2.7 to 5.4] |  |  | 5.4 [3.9 to 6.7] | 5.6 [4.1 to 6.7]
Statistical Analysis 1: Comparison: Dalotuzumab 10 mg/kg Q1W (DB) vs Placebo + Cetuximab + Irinotecan (DB); Test type: Superiority or Other; p = 0.07, Regression, Cox; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [0.98 to 1.83]
Statistical Analysis 2: Comparison: Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (DB) vs Placebo + Cetuximab + Irinotecan (DB); Test type: Superiority or Other; p = 0.44, Regression, Cox; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.83 to 1.55]

3. Primary Outcome: Percentage of Participants Who Have a Clinical or Laboratory Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 to 5 Toxicity
Description: An adverse event (AE) was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure. (Grade 3=Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living. Grade 4=Life-threatening consequences; urgent intervention indicated. Grade 5=Death related to AE.) Participants were monitored for AEs until the earlier of study discontinuation or 30 days after dalotuzumab/placebo discontinuation. AE grades were assessed using the National Cancer Institute (NCI) CTCAE, version 3.0.
Time Frame: Up to 30 days after last dose of study drug (Up to 33 months)
Population: The All Participants as Treated (APaT) population consisted of all randomized participants who received ≥1 dose of study drug. Participants were included in the treatment group corresponding to the study drug they actually received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dalotuzumab 10 mg/kg Q1W (DB) | Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (OL) | Dalotuzumab 10 mg/kg Q1W (OL) | Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (DB) | Placebo + Cetuximab + Irinotecan (DB)
Number analyzed (Participants) | 180 | 8 | 10 | 180 | 178
Percentage of Participants | 82.8 | 100.0 | 90.0 | 81.1 | 75.8

4. Primary Outcome: Percentage of Participants Who Have a Drug-related Clinical or Laboratory CTCAE Grade 3 to 5 Toxicity
Description: An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure. (Grade 3=Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living. Grade 4=Life-threatening consequences; urgent intervention indicated. Grade 5=Death related to AE.) Drug-related AEs were those AEs that were possibly, probably, or definitely related to study drug or protocol-specified procedures. Participants were monitored for AEs related to dalotuzumab or placebo until the earlier of study discontinuation or 30 days after dalotuzumab/placebo discontinuation. AE grades were assessed using the NCI CTCAE, version 3.0.
Time Frame: Up to 30 days after last dose of study drug (Up to 33 months)
Population: The APaT population consisted of all randomized participants who received ≥1 dose of study drug. Participants were included in the treatment group corresponding to the study drug they actually received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dalotuzumab 10 mg/kg Q1W (DB) | Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (OL) | Dalotuzumab 10 mg/kg Q1W (OL) | Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (DB) | Placebo + Cetuximab + Irinotecan (DB)
Number analyzed (Participants) | 180 | 8 | 10 | 180 | 178
Percentage of Participants | 67.8 | 100.0 | 90.0 | 72.8 | 61.8

5. Primary Outcome: Percentage of Participants Who Discontinue Study Drug Due to an AE
Description: An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure. The percentage of participants who discontinued study drug due to an AE is presented.
Time Frame: Up to last dose of study drug (Up to 32 months)
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Dalotuzumab 10 mg/kg Q1W (DB) | Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (OL) | Dalotuzumab 10 mg/kg Q1W (OL) | Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (DB) | Placebo + Cetuximab + Irinotecan (DB)
Number analyzed (Participants) | 180 | 8 | 10 | 180 | 178
Percentage of Participants | 11.1 | 25.0 | 30.0 | 7.2 | 11.8

6. Primary Outcome: Percentage of Participants Who Experience an AE of Infusion Site Reaction
Description: The percentage of participants who experienced an AE of infusion site reaction is presented.
Time Frame: Up to 30 days after last dose of study drug (Up to 33 months)
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Dalotuzumab 10 mg/kg Q1W (DB) | Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (OL) | Dalotuzumab 10 mg/kg Q1W (OL) | Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (DB) | Placebo + Cetuximab + Irinotecan (DB)
Number analyzed (Participants) | 180 | 8 | 10 | 180 | 178
Percentage of Participants | 0.0 | 12.5 | 0.0 | 0.0 | 0.0

7. Secondary Outcome: Overall Response Rate (ORR) of Dalotuzumab in Combination With Cetuximab + Irinotecan Versus ORR of Cetuximab + Irinotecan Alone in Participants With Wild Type of Colorectal Cancer
Description: ORR, using RECIST 1.0, was defined as the percentage of participants in the analysis population who had a confirmed Complete Response (CR; disappearance of all target lesions) or Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions) at any time during the study, based on central radiology review.
Time Frame: Every 6 weeks (Up to 32 months)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Dalotuzumab 10 mg/kg Q1W (DB) | Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (OL) | Dalotuzumab 10 mg/kg Q1W (OL) | Dalotuzumab 15 mg/kg/7.5 mg/kg Q2W (DB) | Placebo + Cetuximab + Irinotecan (DB)
Number analyzed (Participants) | 116 | 0 | 0 | 117 | 111
Percentage of Participants | 21.6 |  |  | 23.9 | 26.1

ADVERSE EVENTS:
Time Frame: Up to 30 days after last dose of study drug (Up to 33 months)
Description: The APaT population consisted of all randomized participants who received ≥1 dose of study drug. Participants were included in the treatment group corresponding to the study drug they actually received.
Groups:
- Dalotuzumab 10 mg/kg Q1W (BD): In DB Week 1, participants received cetuximab 400 mg/m^2 IV loading dose and irinotecan IV at their pre-study dosage. Starting with DB Week 2, participants received cetuximab 250 mg/m^2 IV Q1W maintenance dose, irinotecan IV Q1W and DB dalotuzumab 10 mg/kg IV Q1W for up to 32 months of treatment.
- Dalotuzumab 15 mg/kg /7.5 mg/kg Q2W (OL): In the OL portion of the study, ≥6 participants received cetuximab 400 mg/m^2 Q1W + irinotecan Q1W at their pre-study dosage + OL dalotuzumab (loading dose of 15 mg/kg IV followed by a maintenance dose of 7.5 mg/kg 2 weeks later) to verify the safety of the regimen. In DB Week 1, participants received cetuximab 400 mg/m^2 IV + irinotecan IV. In DB Week 2, participants received cetuximab 250 mg/m^2 IV + irinotecan IV + DB dalotuzumab 15 mg/kg IV. In DB Week 3, participants received cetuximab 250 mg/m^2 IV + irinotecan IV. Starting with DB Week 4, participants received cetuximab 250 mg/m^2 IV Q1W + irinotecan IV Q1W + DB dalotuzumab 7.5 mg/kg IV Q2W for up to 32 months of treatment.
- Dalotuzumab 15 mg/kg /7.5 mg/kg Q2W (DB): In DB Week 1, participants received cetuximab 400 mg/m^2 IV + irinotecan IV at their pre-study dosage. In DB Week 2, participants received cetuximab 250 mg/m^2 IV + irinotecan IV + DB dalotuzumab 15 mg/kg IV. In DB Week 3, participants received cetuximab 250 mg/m^2 IV + irinotecan IV. Starting with DB Week 4, participants received cetuximab 250 mg/m^2 IV Q1W + irinotecan IV Q1W + DB dalotuzumab 7.5 mg/kg IV Q2W for up to 32 months of treatment.
Arm/Group | Dalotuzumab 10 mg/kg Q1W (BD) | Dalotuzumab 15 mg/kg /7.5 mg/kg Q2W (OL) | Dalotuzumab 10 mg/kg Q1W (OL) | Dalotuzumab 15 mg/kg /7.5 mg/kg Q2W (DB) | Placebo + Cetuximab + Irinotecan (DB)
Serious Adverse Events (participants affected / at risk) | 94/180 | 5/8 | 4/10 | 77/180 | 75/178
Other Adverse Events (participants affected / at risk) | 178/180 | 8/8 | 10/10 | 174/180 | 172/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalotuzumab 10 mg/kg Q1W (BD) (N=180) | Dalotuzumab 15 mg/kg /7.5 mg/kg Q2W (OL) (N=8) | Dalotuzumab 10 mg/kg Q1W (OL) (N=10) | Dalotuzumab 15 mg/kg /7.5 mg/kg Q2W (DB) (N=180) | Placebo + Cetuximab + Irinotecan (DB) (N=178)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (6) | 0 (0) | 0 (0) | 7 (8) | 4 (5)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blindness transient (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 13 (13) | 1 (1) | 1 (1) | 10 (14) | 7 (8)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 9 (10)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (3)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (2) | 4 (4) | 3 (3)
Asthenia (General disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 8 (10)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary sepsis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Isosporiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 3 (4)
Pneumonia necrotising (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 34 (34) | 0 (0) | 0 (0) | 27 (27) | 27 (27)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic hyperosmolar coma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postrenal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalotuzumab 10 mg/kg Q1W (BD) (N=180) | Dalotuzumab 15 mg/kg /7.5 mg/kg Q2W (OL) (N=8) | Dalotuzumab 10 mg/kg Q1W (OL) (N=10) | Dalotuzumab 15 mg/kg /7.5 mg/kg Q2W (DB) (N=180) | Placebo + Cetuximab + Irinotecan (DB) (N=178)
Anaemia (Blood and lymphatic system disorders) | 28 (70) | 1 (1) | 0 (0) | 27 (83) | 34 (82)
Leukopenia (Blood and lymphatic system disorders) | 19 (46) | 0 (0) | 2 (2) | 23 (88) | 28 (69)
Lymphopenia (Blood and lymphatic system disorders) | 5 (11) | 0 (0) | 0 (0) | 4 (13) | 15 (20)
Neutropenia (Blood and lymphatic system disorders) | 74 (249) | 0 (0) | 3 (7) | 81 (375) | 75 (317)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (4)
Conjunctivitis (Eye disorders) | 8 (11) | 1 (2) | 1 (1) | 10 (18) | 15 (25)
Dark circles under eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Eye pruritus (Eye disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 5 (6)
Vision blurred (Eye disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 3 (4)
Abdominal discomfort (Gastrointestinal disorders) | 5 (6) | 1 (1) | 0 (0) | 7 (9) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 57 (94) | 3 (3) | 3 (3) | 57 (100) | 65 (141)
Abdominal pain upper (Gastrointestinal disorders) | 11 (19) | 0 (0) | 0 (0) | 12 (15) | 16 (24)
Anal fissure (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (3) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 48 (90) | 2 (2) | 2 (2) | 40 (68) | 48 (79)
Diarrhoea (Gastrointestinal disorders) | 138 (567) | 4 (18) | 9 (37) | 118 (445) | 121 (507)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 11 (13) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 18 (21) | 1 (2) | 1 (2) | 13 (16) | 24 (38)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (7) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 90 (196) | 4 (6) | 5 (7) | 101 (236) | 96 (292)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 10 (11) | 0 (0) | 1 (1) | 7 (8) | 3 (3)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0) | 4 (4) | 7 (7)
Rectal tenesmus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (6) | 0 (0)
Reflux oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 95 (223) | 1 (2) | 6 (9) | 104 (255) | 67 (162)
Vomiting (Gastrointestinal disorders) | 62 (99) | 2 (3) | 1 (2) | 57 (120) | 51 (124)
Asthenia (General disorders) | 48 (145) | 4 (12) | 3 (12) | 55 (156) | 38 (93)
Fatigue (General disorders) | 74 (154) | 3 (8) | 1 (5) | 63 (119) | 60 (161)
Infusion site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 5 (7) | 0 (0) | 1 (1) | 4 (6) | 6 (8)
Mucosal inflammation (General disorders) | 12 (22) | 1 (1) | 1 (1) | 14 (29) | 8 (18)
Oedema peripheral (General disorders) | 11 (14) | 0 (0) | 0 (0) | 10 (15) | 16 (21)
Pyrexia (General disorders) | 18 (22) | 0 (0) | 0 (0) | 13 (15) | 29 (34)
Hyperbilirubinaemia (Hepatobiliary disorders) | 9 (20) | 0 (0) | 1 (1) | 7 (9) | 7 (12)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 6 (6) | 0 (0) | 1 (1) | 9 (10) | 6 (6)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 51 (151) | 2 (5) | 3 (3) | 62 (183) | 37 (91)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Syphilis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 13 (20) | 0 (0) | 2 (2) | 10 (12) | 6 (6)
Vulvovaginal candidiasis (Infections and infestations) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (4) | 0 (0) | 1 (1) | 3 (11) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 32 (80) | 0 (0) | 0 (0) | 24 (70) | 16 (50)
Aspartate aminotransferase increased (Investigations) | 17 (42) | 0 (0) | 0 (0) | 18 (59) | 15 (33)
Blood alkaline phosphatase increased (Investigations) | 7 (11) | 0 (0) | 0 (0) | 7 (8) | 11 (14)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 37 (40) | 0 (0) | 0 (0) | 37 (41) | 20 (25)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 106 (208) | 1 (1) | 3 (5) | 90 (191) | 74 (164)
Dehydration (Metabolism and nutrition disorders) | 6 (11) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 62 (220) | 1 (4) | 3 (9) | 64 (292) | 33 (77)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 13 (27) | 0 (0) | 1 (1) | 11 (20) | 8 (19)
Hypokalaemia (Metabolism and nutrition disorders) | 15 (21) | 1 (2) | 1 (5) | 8 (10) | 15 (19)
Hypomagnesaemia (Metabolism and nutrition disorders) | 37 (163) | 2 (23) | 2 (22) | 43 (131) | 37 (124)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (30) | 1 (1) | 1 (1) | 21 (26) | 15 (34)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 10 (11) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (9) | 2 (4) | 2 (2) | 9 (15) | 7 (11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0) | 0 (0) | 11 (16) | 8 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (12) | 1 (1) | 0 (0) | 8 (10) | 13 (18)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 16 (24) | 0 (0) | 0 (0) | 21 (31) | 21 (25)
Dysgeusia (Nervous system disorders) | 7 (7) | 0 (0) | 2 (2) | 8 (14) | 6 (6)
Headache (Nervous system disorders) | 14 (14) | 0 (0) | 0 (0) | 12 (14) | 15 (39)
Lethargy (Nervous system disorders) | 17 (75) | 0 (0) | 2 (5) | 13 (33) | 19 (90)
Neuropathy peripheral (Nervous system disorders) | 6 (6) | 0 (0) | 0 (0) | 4 (4) | 10 (13)
Peripheral sensory neuropathy (Nervous system disorders) | 11 (25) | 0 (0) | 0 (0) | 15 (36) | 5 (11)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 3 (4) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Depression (Psychiatric disorders) | 3 (4) | 0 (0) | 1 (1) | 4 (4) | 4 (5)
Insomnia (Psychiatric disorders) | 23 (25) | 0 (0) | 0 (0) | 16 (18) | 23 (35)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (31) | 0 (0) | 1 (2) | 29 (47) | 25 (29)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 (28) | 0 (0) | 0 (0) | 22 (28) | 25 (34)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 2 (2) | 3 (5) | 14 (22) | 18 (21)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 1 (1) | 5 (5) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0) | 1 (1) | 9 (9) | 7 (8)
Acne (Skin and subcutaneous tissue disorders) | 11 (35) | 1 (1) | 0 (0) | 23 (48) | 15 (33)
Alopecia (Skin and subcutaneous tissue disorders) | 46 (80) | 2 (3) | 1 (2) | 50 (68) | 50 (70)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 88 (195) | 8 (18) | 9 (31) | 86 (186) | 81 (231)
Dry skin (Skin and subcutaneous tissue disorders) | 59 (95) | 2 (2) | 4 (5) | 64 (96) | 57 (85)
Nail disorder (Skin and subcutaneous tissue disorders) | 8 (24) | 0 (0) | 1 (1) | 15 (35) | 6 (13)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 16 (29) | 1 (1) | 2 (5) | 15 (29) | 12 (25)
Pruritus (Skin and subcutaneous tissue disorders) | 43 (69) | 1 (1) | 3 (3) | 53 (93) | 43 (77)
Rash (Skin and subcutaneous tissue disorders) | 76 (217) | 0 (0) | 0 (0) | 66 (184) | 60 (165)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (5) | 0 (0) | 4 (5) | 6 (6)
Skin fissures (Skin and subcutaneous tissue disorders) | 47 (86) | 2 (2) | 1 (1) | 55 (108) | 48 (105)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 7 (13) | 0 (0) | 0 (0) | 10 (24) | 4 (10)
Flushing (Vascular disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 3 (5)
Hypertension (Vascular disorders) | 3 (4) | 2 (2) | 0 (0) | 2 (2) | 8 (14)
Hypotension (Vascular disorders) | 3 (4) | 1 (1) | 0 (0) | 4 (6) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.